CLINICAL TRIAL: NCT05359185
Title: Empowering Families Project: An RCT of the Effects of Relationship Education With and Without Ancillary Economic Services on Family Outcomes
Brief Title: Empowering Families Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Principal Investigator, Hannah Williamson, Associate Professor, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 90ZB0025
Record Dates: First submitted 2022-04-27; First posted 2022-05-03 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Couples; Relationship, Marital; Relational Problems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment-only (Experimental): Participants in the this group will receive core Relationship Education programming, which consists of six weekly 2.5-hour Family Wellness Workshops.
  Interventions: Behavioral: Family Wellness
- Treatment-Plus (Experimental): Participants in this group will receive an enhanced model that includes the core RE programming, and adds economic-focused services which include two 2.5-hour workshops (one on financial planning and one on career coaching), as well as individual financial planning and career coaching services ongoing for up to one year.
  Interventions: Behavioral: Family Wellness; Behavioral: Career Coaching; Behavioral: Financial Planning

INTERVENTIONS:
Behavioral: Family Wellness — https://familywellness.com/
Behavioral: Career Coaching — Individualized career coaching and employment services.
  Arms: Treatment-Plus
Behavioral: Financial Planning — Individualized financial planning services.
  Arms: Treatment-Plus

SUMMARY:
This RCT will test the marginal benefit of adding economic-focused services to traditional relationship education (RE) interventions. 344 couples will be randomly assigned to the RE only or RE plus economic-services condition. All couples will be assessed at baseline, 6-weeks, 6-months, and 12-months. This project will examine whether couples in the RE plus condition have better relationship and economic outcomes than couples in the RE only condition.

ELIGIBILITY:
Inclusion Criteria:

* couples involved in a romantic relationship

Exclusion Criteria:

* current domestic violence or child maltreatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 666 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2025-09-29 (Actual); Study Completion 2025-09-29 (Actual)

PRIMARY OUTCOMES:
Change in Relationship satisfaction | From baseline to 6-weeks, 6-months, 12-months
  Couples Satisfaction Index (CSI-4).
Changes in Positive Communication | From baseline to 6-weeks, 6-months, 12-months
  Seven items, scored on four-point scale and averaged. Sample item: "My partner and I were good at working out our differences."
Changes in Negative Communication | From baseline to 6-weeks, 6-months, 12-months
  Nine items, scored on four-point scale and averaged. Sample item: "My partner was rude or mean to me when we disagree."
Changes in Income | From baseline to 6-months, 12-months
  Single item: "How much would you say you personally as an individual earned in total from all work in the last month, before taxes and deductions?" Open numeric response
Changes in Financial Strain | From baseline to 6-months, 12-months
  Five items assess the degree of difficulty the household has had fulfilling financial obligations and purchasing necessary items. Items scored on a 4-point scale and averaged.
Changes in Financial Capability | From baseline to 6-months, 12-months
  Six items assess capability to manage household finances, (e.g., "In the last 2 months, have you been charged a late fee on a loan or bill?"). Items summed to form an index with range of 0-8 (two 3-point items, four 2-point items.

SECONDARY OUTCOMES:
Changes in Support and Affection | From baseline to 6-weeks, 6-months, 12-months
  Five items, scored on four-point scale and averaged. Sample item: "My partner knows and understands me."
Changes in Wealth | From baseline to 6-months, 12-months
  Single item: "About how much money does your household have saved somewhere (in a savings account, 401k, hidden cash envelope, etc.)?" Open numeric response

CONTACTS AND LOCATIONS:
Locations (1):
- The Parenting Center, Fort Worth, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
Fully de-identified datasets may be shared with other researchers in the future.

DOCUMENTS (1):
  • Statistical Analysis Plan (2022-04-27): https://cdn.clinicaltrials.gov/large-docs/85/NCT05359185/SAP_000.pdf